CLINICAL TRIAL: NCT02755233
Title: Ipilimumab-induced Lung Toxicity: A Prospective Observational Study on Pulmonary Function Changes in Patients With Metastatic Melanoma
Brief Title: Ipilimumab-induced Lung Toxicity: Observational Study
Acronym: Ipi-Lu-Tox
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0191
Record Dates: First submitted 2016-04-15; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary function: Patients in whom treatment with ipilimumab due to metastatic melanoma is indicated
  Interventions: Other: Pulmonary Function

INTERVENTIONS:
Other: Pulmonary Function — Spirometry and DLCO were measured according to performance standards based on the statements from the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Values of DLCO were adjusted for the patient's current hemoglobin value, and the patients were asked to withhold cigarette smoking at least four hours before pulmonary function testing. Lung volumes and DLCO were measured with a commercial ZAN300 CO Diffusion system (nSpire Health GmbH, Oberthulba, Germany)
  Other Names: Spirometry and CO-diffusion capacity measurement

SUMMARY:
Serial spirometries and measurements of CO-diffusion capacity (DLCO) in patients with MM before and during treatment with ipilimumab are performed. A reduction from baseline of forced vital capacity (FVC) of ≥10%, or ≥15% of DLCO was defined clinically meaningful, thus indicative for pulmonary toxicity.

DETAILED DESCRIPTION:
The aim of this prospective observational study is to determine the prevalence of ipilimumab lung toxicity defined by a significant decline of the diffusing capacity of the lung for carbon monoxide (DLCO) and/or forced vital capacity (FVC) in patients with MM.

Patients aged over 18 years with an established diagnosis of MM who are treated and followed up at the Department of Dermatology are asked to participate in the study after the indication for treatment with ipilimumab is given by the interdisciplinary skin tumorboard conference. After written informed consent is obtained, patients undergo a baseline evaluation (V1) including a medical history, physical examination, laboratory analyses (hemoglobin, leucocytes count, C-reactive protein, and pulmonary function tests (PFTs) with spirometry and measurement of DLCO. Thereafter, the first dose of ipilimumab (3mg/kg) is given intravenously over a period of 90 minutes without premedication. The subsequent three doses of ipilimumab are administered three weekly with analogue dose. Subsequent study visits (V2, V3, V4) including PFTs are scheduled on the same day as ipilimumab is administered. Thus, study visits are thoroughly adapted to the clinical visits, which is given by the administration of ipilimumab (total of four injections each separated by three weeks). In case of new respiratory symptoms during the study period, additional PFTs and a high-resolution computed tomography (HR-CT) of the chest are performed. In case of early study termination during follow-up pulmonary function test values which are already obtained are used for the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of metastatic melanoma

Exclusion Criteria:

* Acute pulmonary infection at enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom a treatment with ipilimumab due to metastatic melanoma is indicated
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Relative reduction of DLCO of more than 15% from the baseline value during follow-up | 9 weeks
  A relative reduction of ≥15% from baseline of DLCO was chosen as clinically meaningful, thus indicative of a possible interstitial lung disease as a consequence of ipilimumab induced pulmonary toxicity

SECONDARY OUTCOMES:
Relative reduction of FVC of more than 10% from the baseline value during | 9 weeks
  A relative reduction of FVC of ≥10% from baseline was chosen as clinically meaningful, thus indicative of a possible interstitial lung disease as a consequence of ipilimumab induced pulmonary toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Divison of Pneumology
Locations (1):
- Department of Pulmonology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Additional supporting file